CLINICAL TRIAL: NCT02613871
Title: A Phase 3b Open-Label Study of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 1 or 2 Hepatitis C Virus (HCV) and Hepatitis B Virus (HBV) Coinfection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed-Dose Combination in Adults With Chronic HCV and HBV Coinfection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1655
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LDV/SOF (Experimental): LDV/SOF FDC for 12 weeks
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to determine the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in adults with chronic genotype 1 or 2 HCV infection who are coinfected with HBV in Taiwan.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals ≥ 40 kg in weight with chronic genotype 1 or 2 HCV and HBV coinfection
* Individuals must not be taking or requiring treatment with HBV antiviral therapy at screening. For participants that are HBV treatment experienced, the most recent treatment must have been completed at least 6 months prior to Day 1.
* Cirrhosis determination by Fibroscan
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female or male is of childbearing potential

Key Exclusion Criteria:

* Current or prior history of clinically-significant illness or any other major medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol
* Pregnant or nursing female
* Infection with human immunodeficiency virus (HIV) or hepatitis delta virus (HDV)
* Hepatocellular carcinoma (HCC) or other malignancy
* Current or prior history of clinical hepatic decompensation

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- Taiwan (8):
  - Changhua
  - Chiayi City
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Liu CJ, Chuang WL, Sheen IS, Wang HY, Chen CY, Tseng KC, et al. Ledipasvir/Sofosbuvir for 12 Weeks Is Safe and Effective in Patients With Chronic Hepatitis C and Hepatitis B Coinfection: a Phase 3 Study in Taiwan [Poster SAT-243]. EASL: The International Liver Congress; 2019 10-14 April; Vienna, Austria.
- [Result] Liu CJ, Chuang WL, Sheen IS, Wang HY, Chen CY, Tseng KC, et al. Declines in HBsAg Levels Observed During Treatment With Ledispavir/Sofosbuvir in Patients With Chronic Hepatitis B Virus and Hepatitis C Virus Infection [Poster 1083]. The Liver Meeting® 2017 - The 68th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2017 20-24 October; Washington, D. C.
- [Result] Liu CJ, Chuang WL, Sheen IS, Wang HY, Chen CY, Tseng KC, Chang TT, Massetto B, Yang JC, Yun C, Knox SJ, Osinusi A, Camus G, Jiang D, Brainard DM, McHutchison JG, Hu TH, Hsu YC, Lo GH, Chu CJ, Chen JJ, Peng CY, Chien RN, Chen PJ. Efficacy of Ledipasvir and Sofosbuvir Treatment of HCV Infection in Patients Coinfected With HBV. Gastroenterology. 2018 Mar;154(4):989-997. doi: 10.1053/j.gastro.2017.11.011. Epub 2017 Nov 22. PMID 29174546
- [Result] Liu CJ, Chuang WL, Sheen IS, Wang HY, Chen CY, Tseng KC, et al. Ledipasvir/Sofosbuvir for 12 Weeks Is Safe and Effective in Patients with Chronic Hepatitis C and Hepatitis B Coinfection: A Phase 3 Study in Taiwan [Presentation]. The International Liver Congress™ 2017: European Association for the Study of the Liver (EASL); 2017 19-23 April; Amsterdam, the Netherlands.
- [Derived] Liu CJ, Sheen IS, Chen CY, Chuang WL, Wang HY, Tseng KC, Chang TT, Yang J, Massetto B, Suri V, Camus G, Jiang D, Zhang F, Gaggar A, Hu TH, Hsu YC, Lo GH, Chu CJ, Chen JJ, Peng CY, Chien RN, Chen PJ. Ledipasvir/Sofosbuvir for Patients Coinfected With Chronic Hepatitis C and Hepatitis B in Taiwan: Follow-up at 108 Weeks Posttreatment. Clin Infect Dis. 2022 Aug 31;75(3):453-459. doi: 10.1093/cid/ciab971. PMID 34864948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Taiwan. The first participant was screened on 22 December 2015. The last study visit occurred on 07 November 2018.
Pre-assignment Details: 135 participants were screened.
Groups:
- LDV/SOF FDC: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | LDV/SOF FDC
Started | 111
Completed | 108
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Groups:
- LDV/SOF FDC: LDV/SOF (90/400 mg) FDC tablet orally once daily for 12 weeks.
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 99
  Ethnicity: Not Permitted | 12
IL28b Status [Count of Participants; unit: Participants] — CC and CT alleles are different forms of the IL28b gene.
  Participants
    CC | 85
    CT | 26
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.73)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 44
  ≥ 800,000 IU/mL | 67
Cirrhosis status [Count of Participants; unit: Participants]
  Absence | 93
  Presence | 18
Fibroscan Score [Mean (Standard Deviation); unit: kPa] — FibroScan® is a non-invasive device that assesses the hardness (or stiffness) of the liver using the technique of transient elastography. FibroScan results range from 2.5 kPa to 75 kPa with higher scores indicating greater liver stiffness. Per protocol, cirrhosis status was determined as follows:
  * Presence of cirrhosis = FibroScan® result of > 12.5 kPa
  * Absence of cirrhosis = FibroScan® result of ≤ 12.5 kPa
  kPa | 9.3 (7.05)
Hepatitis B Virus (HBV) DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 2.1 (0.92)
Plasma HBV DNA [Mean (Standard Deviation); unit: IU/mL] | 9423.1 (69641.90)
HBsAg [Mean (Standard Deviation); unit: IU/mL] | 578.6 (1113.56)
Serum Lysyl Oxidase-Like 2 (LOXL-2) Level [Mean (Standard Deviation); unit: pg/mL] | 98 (64.4)
HCV Genotype [Count of Participants; unit: Participants] — HCV Genotype 1 indicates genotype 1 with no confirmed subtype (eg, 1a, 1b or mixed 1a/1b).
  Participants
    Genotype 1 | 1
    Genotype 1a | 3
    Genotype 1b | 64
    Genotype 2 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantification (LLOQ; 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants
  Genotype 1: number analyzed (Participants) | 68
  Genotype 1 | 100.0 [94.7 to 100.0]
  Genotype 2: number analyzed (Participants) | 43
  Genotype 2 | 100.0 [91.8 to 100.0]
  Total | 100.0 [96.7 to 100.0]

2. Primary Outcome: Percentage of Participants With Any Adverse Event Leading to Permanent Discontinuation of Study Drug
Time Frame: First dose date up to 12 weeks
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants | 0.0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ (15 IU/mL) at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants | 100.0 [96.7 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment
Description: LLOQ = 15 IU/mL
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants
  Week 1 | 33.3 [24.7 to 42.9]
  Week 2 | 82.0 [73.6 to 88.6]
  Week 4 | 100.0 [96.7 to 100.0]
  Week 8 | 100.0 [96.7 to 100.0]
  Week 12 | 100.0 [96.7 to 100.0]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Posttreatment Weeks 24, 36, 48, 60, 72, 84, 96, and 108
Description: LLOQ = 15 IU/mL
Time Frame: Posttreatment Weeks 24, 36, 48, 60, 72, 84, 96, and 108
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants
  Posttreatment Week 24 | 100 [96.7 to 100]
  Posttreatment Week 36 | 100 [96.7 to 100]
  Posttreatment Week 48 | 100 [96.7 to 100]
  Posttreatment Week 60 | 100 [96.7 to 100]
  Posttreatment Week 72: number analyzed (Participants) | 110
  Posttreatment Week 72 | 100 [96.7 to 100]
  Posttreatment Week 84: number analyzed (Participants) | 109
  Posttreatment Week 84 | 100 [96.7 to 100]
  Posttreatment Week 96: number analyzed (Participants) | 108
  Posttreatment Week 96 | 100 [96.6 to 100]
  Posttreatment Week 108: number analyzed (Participants) | 108
  Posttreatment Week 108 | 100 [96.6 to 100]

6. Secondary Outcome: HCV RNA Change From Baseline While on Treatment
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Week 1 | -4.14 (0.551)
  Change at Week 2 | -4.63 (0.702)
  Change at Week 4 | -4.73 (0.727)
  Change at Week 8 | -4.73 (0.727)
  Change at Week 12 | -4.73 (0.727)

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as :
  * Breakthrough (confirmed HCV RNA ≥ LLOQ [15 IU/mL] after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment), or
  * Relapse (HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement)
Time Frame: First dose date up to Posttreatment Week 12
Population: Participants in Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants | 0

8. Secondary Outcome: Plasma HBV DNA Change From Baseline While on Treatment
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Week 1 | -0.06 (0.237)
  Change at Week 2 | 0.08 (0.366)
  Change at Week 4 | 0.37 (0.705)
  Change at Week 8 | 0.51 (0.906)
  Change at Week 12: number analyzed (Participants) | 106
  Change at Week 12 | 0.24 (0.746)

9. Secondary Outcome: Plasma HBV DNA Change From Baseline at Posttreatment Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, and 108
Time Frame: Posttreatment Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, and 108
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Posttreatment Week 4 | 0.49 (0.727)
  Change at Posttreatment Week 12 | 0.66 (0.955)
  Change at Posttreatment Week 24 | 0.56 (1.036)
  Change at Posttreatment Week 36 | 0.67 (1.190)
  Change at Posttreatment Week 48 | 0.68 (1.269)
  Change at Posttreatment Week 60 | 0.70 (1.399)
  Change at Posttreatment Week 72: number analyzed (Participants) | 110
  Change at Posttreatment Week 72 | 0.55 (1.131)
  Change at Posttreatment Week 84: number analyzed (Participants) | 109
  Change at Posttreatment Week 84 | 0.50 (1.008)
  Change at Posttreatment Week 96: number analyzed (Participants) | 108
  Change at Posttreatment Week 96 | 0.41 (0.963)
  Change at Posttreatment Week 108: number analyzed (Participants) | 108
  Change at Posttreatment Week 108 | 0.38 (0.923)

10. Secondary Outcome: HBsAg Level Change From Baseline While on Treatment
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Week 1 | -0.14 (0.184)
  Change at Week 2 | -0.18 (0.181)
  Change at Week 4 | -0.25 (0.185)
  Change at Week 8 | -0.41 (0.234)
  Change at Week 12: number analyzed (Participants) | 106
  Change at Week 12 | -0.47 (0.266)

11. Secondary Outcome: HBsAg Level Change From Baseline at Posttreatment Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, and 108
Time Frame: Posttreatment Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, and 108
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Posttreatment Week 4 | -0.16 (0.347)
  Change at Posttreatment Week 12 | -0.01 (0.338)
  Change at Posttreatment Week 24 | -0.02 (0.405)
  Change at Posttreatment Week 36 | -0.07 (0.484)
  Change at Posttreatment Week 48 | -0.10 (0.526)
  Change at Posttreatment Week 60 | -0.16 (0.664)
  Change at Posttreatment Week 72: number analyzed (Participants) | 110
  Change at Posttreatment Week 72 | -0.20 (0.619)
  Change at Posttreatment Week 84: number analyzed (Participants) | 109
  Change at Posttreatment Week 84 | -0.25 (0.608)
  Change at Posttreatment Week 96: number analyzed (Participants) | 108
  Change at Posttreatment Week 96 | -0.32 (0.618)
  Change at Posttreatment Week 108: number analyzed (Participants) | 108
  Change at Posttreatment Week 108 | -0.37 (0.658)

12. Secondary Outcome: Serum LOXL-2 Level Change From Baseline While on Treatment
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
pg/mL
  Change at Week 1: number analyzed (Participants) | 110
  Change at Week 1 | -2 (29.4)
  Change at Week 2 | -6 (26.9)
  Change at Week 4 | -15 (27.8)
  Change at Week 8 | -22 (36.6)
  Change at Week 12: number analyzed (Participants) | 106
  Change at Week 12 | -27 (36.0)

13. Secondary Outcome: Serum LOXL-2 Level Change From Baseline at Posttreatment Weeks 4, 12, and 36
Time Frame: Posttreatment Weeks 4, 12, and 36
Population: Participants in Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
pg/mL
  Change at Posttreatment Week 4 | -30 (45.0)
  Change at Posttreatment Week 12 | -32 (51.8)
  Change at Posttreatment Week 36 | -41 (53.0)

14. Secondary Outcome: Percentage of Participants That Required HBV Therapy During the Study
Time Frame: First dose date up to Posttreatment Week 108
Population: Participants in Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants | 7.2

15. Secondary Outcome: Fibrosis Status as Assessed by Fibroscan Score at Posttreatment Weeks 12, 60, and 108
Description: FibroScan is a non-invasive device that assesses the hardness (or stiffness) of the liver using the technique of transient elastography. FibroScan results range from 2.5 kPa to 75 kPa with higher scores indicating greater liver stiffness. Per protocol, cirrhosis status was determined as follows:
  * Presence of cirrhosis = FibroScan result of > 12.5 kPa
  * Absence of cirrhosis = FibroScan result of ≤ 12.5 kPa
Time Frame: Posttreatment Weeks 12, 60, and 108
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
kPa
  Posttreatment Week 12 | 8.0 (7.01)
  Posttreatment Week 60 | 7.2 (4.99)
  Posttreatment Week 108: number analyzed (Participants) | 108
  Posttreatment Week 108 | 7.1 (4.79)

16. Secondary Outcome: Percentage of Participants That Develop Hepatocellular Carcinoma (HCC) During the Study
Time Frame: First dose date up to Posttreatment Week 108
Population: Participants in Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF FDC
Number analyzed (Participants) | 111
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 12 weeks plus 30 days; All-Cause Mortality: First dose date up to maximum 3 years
Description: Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | LDV/SOF FDC
All-Cause Mortality (participants affected / at risk) | 2/111
Serious Adverse Events (participants affected / at risk) | 4/111
Other Adverse Events (participants affected / at risk) | 24/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF FDC (N=111)
Duodenal ulcer (Gastrointestinal disorders) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Optic neuritis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF FDC (N=111)
Fatigue (General disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 9
Headache (Nervous system disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years